CLINICAL TRIAL: NCT02569827
Title: A Phase Ib/IIa Single Centre, Double-blind, Double-dummy, Placebo-controlled, Parallel-group Dose Ranging Trial in Adult Participants With Uncomplicated Dengue Fever in Singapore
Brief Title: Celgosivir or Modipafant as Treatment for Adult Participants With Uncomplicated Dengue Fever in Singapore
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The investigational drug celgosivir will not be developed due to lack of VC funding.
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); 60 Degrees Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cel01
Record Dates: First submitted 2015-10-01; First posted 2015-10-07 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Dengue Fever
Keywords: Uncomplicated Dengue Fever; Treatment; Phase Ib/IIa; single centre; double-blind; placebo-controlled; parallel-group dose ranging trial; Modipafant; Celgosivir
MeSH Terms: conditions — Dengue | interventions — celgosivir; modipafant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Placebo Comparator): Placebo Q6H for 5 days
  A total of 72 participants (18 participants per group assuming up to two drop-outs per group) will be assigned in a randomised double-blind fashion.
  Interventions: Drug: Placebo
- Cohort 2 (Active Comparator): Modipafant 50 mg Q12H alternating with placebo Q12H for 5 days (total of 10 modipafant doses = 500 mg)
  Interventions: Drug: Modipafant 50mg
- Cohort 3 (Active Comparator): Modipafant 100 mg Q12H alternating with placebo Q12H 5 days (total of 10 modipafant doses = 1000 mg)
  Interventions: Drug: Modipafant 100mg
- Cohort 4 (Active Comparator): Celgosivir 150 mg Q6H for 5 days (total of 20 doses = 3000 mg total).
  Interventions: Drug: Celgosivir

INTERVENTIONS:
Drug: Celgosivir — Celgosivir 150 mg Q6H for 5 days (total of 20 doses = 3000 mg celgosivir total).
  Arms: Cohort 4
Drug: Modipafant 50mg — Modipafant 50 mg Q12H alternating with placebo Q12H for 5 days (total of 10 modipafant doses = 500 mg modipafant)
  Arms: Cohort 2
Drug: Placebo — Placebo Q6H for 5 days
  Arms: Cohort 1
Drug: Modipafant 100mg — Modipafant 100 mg Q12H alternating with placebo Q12H for 5 days (total of modipafant 10 doses = 1000 mg modipafant)
  Arms: Cohort 3

SUMMARY:
Dengue fever is an acute febrile illness transmitted by mosquitoes, which affects half the world's population. There are 96 million symptomatic infections, 500,0000 hospitalisations and 25,000 deaths per year attributed to the disease. The economic burden is $12 billion. In Singapore, as elsewhere, the incidence of the disease continues to increase despite aggressive control measures. At present there are no approved medicines for treating dengue fever. Only supportive fluid replacement therapy is used to treat vascular leakage in patients with severe illness. Therefore there is an urgent need to find alternative treatments. Experiments in the laboratory have shown that Celgosivir and modipafant inhibit dengue virus and improve mouse survival. Both drugs have previously been used in humans with good safety records, so investigators are taking this one step further to find out how well it works in dengue patients. Investigators plan to enroll dengue patients within 48 hours of fever onset and assign them to one of four treatment groups over five days. Together with the support from the industry partner, 60°Pharmaceuticals PLC, the investigators will determine the safety and effectiveness of these drugs on acute dengue patients and pave the way forward for dengue antiviral medicines to reach patients.

DETAILED DESCRIPTION:
This trial is a single centre, double-blind, double-dummy, placebo-controlled parallel-group, dose ranging study in adult participants with uncomplicated dengue fever. The study will be conducted in two parts:

In Part 1, 72 otherwise healthy participants (18 participants per group, assuming up to 2 dropouts per group) with uncomplicated dengue fever meeting the inclusion/exclusion criteria will be randomised to receive treatment with placebo, celgosivir or modipafant. Participants will be randomised in parallel to one of Cohorts 1 to 4:

* Cohort 1: Placebo Q6Hours for 5 days
* Cohort 2: Modipafant 50 mg Q12Hours alternating with placebo Q12Hours for 5 days (total of 10 modipafant doses = 500 mg);
* Cohort 3: Modipafant 100 mg Q12Hours alternating with placebo Q12Hours 5 days (total of 10 modipafant doses = 1000 mg);
* Cohort 4: Celgosivir 150 mg Q6H for 5 days (total of 20 doses = 3000 mg total).

As modipafant is untested in uncomplicated dengue fever patients, a double-blinded sentinel group consisting of 4 participants randomised in a 1:1:1:1 ratio of Cohort 1: Cohort 2: Cohort 3: Cohort 4 will complete treatment to Study Day 5 prior to continuing enrolment of the remaining participants. Remaining 68 participants will be enrolled in parallel in a double-blinded fashion.

Participants will be evaluated during screening (< 24 hours before Study Day 1) and on Study Days 1-5, 14 and 28. Participants will be confined in the SingHealth Investigational Medicine Unit (IMU) from screening until end of study assessments on Study Day 5 and return to the clinic at Day 14 and 28 as outpatients. All patients will receive capsules Q6H for 5 days prepared by an open-label pharmacist according to the randomisation plan.

Interim Analysis: The treatment regimen chosen for Part 2 will be based on the analysis of Part 1 data. A detailed Statistical Analysis Plan (SAP) will be prepared for approval by the Sponsor prior to performing any unblinded analysis for presentation to personnel designated as being blinded to the randomization. A data safety monitoring board (DSMB) will conduct a blinded review of source verified safety data. If there are no safety concerns, an independent statistician will perform an unblinded futility analysis of preliminary efficacy data from the four cohorts; blinding to treatment group (celgosivir or modipafant) will be maintained, however placebo will be unblinded. If futility is concluded, the Sponsor may elect to discontinue the study. If a signal is detected, a sample size calculation will be undertaken for Part 2. The Sponsor will convene a Scientific Advisory Board (SAB) who will then review unblinded log10 serum viral load AUC for viraemia and platelet count data to recommend which dosing monotherapy dosing regimen to advance to Part 2. If the recommended sample size for Part 2 exceeds the maximum specified for Part 1 and 2 (a total combined sample size of N = 132 participants) for a monotherapy, the Sponsor will submit a major amendment for Institutional Review Board/ Health Science Authority (IRB/HSA) consideration prior to initiating Part 2.

For Part 2, up to 60 otherwise healthy participants with uncomplicated dengue fever meeting the inclusion/exclusion criteria will be assigned in a randomised double-blind fashion to:

* Cohort 5: (i) celgosivir monotherapy 150 mg Q6H, OR (ii) modipafant monotherapy (either 50 mg Q12H or 100 mg Q12H)
* Cohort 6: Placebo extension for 5 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 21-65 years;
2. Acute febrile illness with two or more manifestations (headache, retro-orbital pain, myalgia, arthralgia, rash, haemorrhagic manifestations, or leucopoenia) and occurrence at the same location and time as other confirmed cases of dengue fever;
3. Fever (> 37.5°C) or history of fever at screening
4. < 48 hours of fever history
5. Positive NS1 strip assay or reverse-transcriptase polymerase chain reaction (RT-PCR).
6. Able and willing to give written informed consent; and,
7. Willing to be an inpatient from Study Screening to Study Day 5 and to return to hospital on study Days 14 and 28.
8. Willing to keep a study diary from Study Day 5 to Day 14.

Exclusion Criteria:

1. Clinical signs and symptoms for severe dengue, such as:

   * Severe abdominal pain;
   * Persistent vomiting;
   * CS fluid accumulation;
   * Mucosal bleeding;
   * Altered mental state;
   * Liver enlargement > 2 cm;
   * Systolic blood pressure < 90 mmHg; and
   * Pulse pressure < 20 mmHg.
2. A person with any of the following laboratory values:

   * Haematocrit >52% males; >46% females;
   * Aspartate or alanine aminotransferase (AST or ALT) > 1000 U/L;
   * Room air oxygen saturation < 95%;
   * Absolute neutrophil count < 1500/µL;
   * Platelet count < 80,000/mm3;
   * Creatinine > 165 µmol/L males; > 130 µmol/L females;
   * Haemoglobin < 13.0 g/dL males; < 11.0 g/dL females;
   * Total bilirubin > 24 µmol/L; and
   * Serum CPK > 600 U/L.
3. History of or presently active intestinal disorders such as peptic ulcers, intestinal ulcers, intestinal obstructions, intestinal hernias, ulcerative colitis, malabsorption syndrome, celiac disease, Roemheld's syndrome (gastroesophageal regurgitation disease) or Crohn's disease;
4. Severe diarrhoea (grade 2 or higher according to NIH clinical trial guidelines);
5. Current usage of any anticoagulant drugs including, but not limited to, aspirin, warfarin or clopidogrel;
6. Any other CS acute illness within seven days prior to first study drug administration;
7. History of adverse reactions to celgosivir, castanospermine, modipafant or formulation excipients or history of severe drug or food allergies;
8. Exposure to any new investigational drug within 30 days prior to the study drug administration;
9. CS abnormal physical examination unrelated to dengue infection, chest X-ray or 12-lead ECG at screening such as QTc prolongation (> 450 msec);
10. Women of child bearing potential (WOCBP) who are pregnant, breast feeding or unwilling to avoid pregnancy by the use of highly effective contraception (<1% failure rate per year) including oral and subcutaneous implantable hormonal contraceptives, condoms, diaphragm, or intra-uterine system (IUS), during the period that the experimental drug is administered. Prospective WOCBP must have a negative pregnancy test (point of care).
11. Male participants unwilling to comply with the contraceptive requirements of the study as detailed in Section 4.7 (i.e. abstinence, effective barrier contraception during the study and for 65 days after the last dose of study drug).
12. Current significant medical condition or illness including cardiac arrhythmias, cardiomyopathy or other cardiac disease, asthma or other respiratory disease, diabetes mellitus, renal or hepatic impairment, thyroid disease, Parkinson's disease, epilepsy or history of unexplained blackouts, immunocompromised state including known HIV infection, or any other illness that the Investigator considers should exclude the patient, especially those that require continuation of other medications likely to have an interaction with the study drug.
13. Any condition that would render the informed consent invalid, or limit the ability of the participant to comply with the study requirements.
14. Any condition that, in the opinion of the Investigator, would complicate or compromise the study or well-being of the participant.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Viral load AUC for viremia | Day 1 to Day 5
  Area under the curve (AUC) for serum viral load from baseline to Study Day 5 of Celgosivir dosing
Platelet nadir | Day 1 to Day 5
  Lowest platelet count recorded from baseline to Study Day 5 of Modipafant dosing

SECONDARY OUTCOMES:
Fever clearance time (days) | Day 1 to 28
  The time from the start of treatment to the start of the first 24-hour period during which the tympanic or oral temperature remains below 37.5°C
Duration of illness | Day 1 to 28
  A 24-hour reduction in duration of illness that is treatment related is deemed clinically relevant. Draft criteria to support this include: Absence of fever (< 37.4˚C) for at least 24 hours
Maximum percentage haemoconcentration | Day 1 to 28
  Determined by comparison of the maximum haematocrit detected in the acute phase as compared to baseline
Time to NS1 clearance | Day 1 to 28

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Low, Dr, Principal Investigator — Singapore General Hospital
Locations (1):
- Singhealth Investigational Medicine Unit, Singapore, Singapore

REFERENCES:
- [Background] Low JG, Sung C, Wijaya L, Wei Y, Rathore APS, Watanabe S, Tan BH, Toh L, Chua LT, Hou Y, Chow A, Howe S, Chan WK, Tan KH, Chung JS, Cherng BP, Lye DC, Tambayah PA, Ng LC, Connolly J, Hibberd ML, Leo YS, Cheung YB, Ooi EE, Vasudevan SG. Efficacy and safety of celgosivir in patients with dengue fever (CELADEN): a phase 1b, randomised, double-blind, placebo-controlled, proof-of-concept trial. Lancet Infect Dis. 2014 Aug;14(8):706-715. doi: 10.1016/S1473-3099(14)70730-3. Epub 2014 May 28. PMID 24877997
- [Background] Rathore AP, Paradkar PN, Watanabe S, Tan KH, Sung C, Connolly JE, Low J, Ooi EE, Vasudevan SG. Celgosivir treatment misfolds dengue virus NS1 protein, induces cellular pro-survival genes and protects against lethal challenge mouse model. Antiviral Res. 2011 Dec;92(3):453-60. doi: 10.1016/j.antiviral.2011.10.002. Epub 2011 Oct 12. PMID 22020302
- [Background] Watanabe S, Rathore AP, Sung C, Lu F, Khoo YM, Connolly J, Low J, Ooi EE, Lee HS, Vasudevan SG. Dose- and schedule-dependent protective efficacy of celgosivir in a lethal mouse model for dengue virus infection informs dosing regimen for a proof of concept clinical trial. Antiviral Res. 2012 Oct;96(1):32-5. doi: 10.1016/j.antiviral.2012.07.008. Epub 2012 Jul 31. PMID 22867971
- [Background] Whitby K, Pierson TC, Geiss B, Lane K, Engle M, Zhou Y, Doms RW, Diamond MS. Castanospermine, a potent inhibitor of dengue virus infection in vitro and in vivo. J Virol. 2005 Jul;79(14):8698-706. doi: 10.1128/JVI.79.14.8698-8706.2005. PMID 15994763
- [Derived] Watanabe S, Chan KW, Dow G, Ooi EE, Low JG, Vasudevan SG. Optimizing celgosivir therapy in mouse models of dengue virus infection of serotypes 1 and 2: The search for a window for potential therapeutic efficacy. Antiviral Res. 2016 Mar;127:10-9. doi: 10.1016/j.antiviral.2015.12.008. Epub 2016 Jan 13. PMID 26794905